CLINICAL TRIAL: NCT01795417
Title: Safety and Efficacy of Non-invasive Dermatologic Procedure With XP200 Radiofrequency for the Primary Treatment of Wrinkles and Rhytids
Brief Title: Safety and Efficacy of XP200 Radiofrequency Treatment of Wrinkles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BTL Industries Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XP200 3.25 MHZ RF
Record Dates: First submitted 2013-02-18; First posted 2013-02-20 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2013-08

CONDITIONS: Periorbital Wrinkles
Keywords: wrinkles; rhytids; periorbital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- XP200 device RF treatments (Experimental): Every subject in the study will undergo 4 treatments and will be followed up for 6 months with photoraphic 3 evaluations: before treatment, 3 and 6 months follow-up. Photographs will be scored on a Fitzpatrick scale by 3 blinded evaluators.
  Interventions: Device: RF XP200; Device: XP200 RF device

INTERVENTIONS:
Device: RF XP200 — Four weekly non-invasive periorbital wrinkles treatment with RF XP200 device
Device: XP200 RF device — 4 RF treatments of periorbital region on one side of the face

SUMMARY:
To evaluate the wrinkle-reducing effects of 3.25-MHz radiofrequency (RF) energy delivered in 4 weekly applications to human periorbital skin area by grating pre- and 90-days post treatment photographs on the Fitzpatrick Wrinkle Severity Scale (FWSS) by three blinded evaluators.

ELIGIBILITY:
Inclusion Criteria:

* 35-60 years old
* periorbital wrinkles

Exclusion Criteria:

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2012-08; Primary Completion 2012-12 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Improvement in wrinkles appearance | 3 months
  One point or greater improvement in periorbital wrinkle score on a Fitzpatrick scale 3 months after last treatment as determined by at least 2 out of 3 blinded photographs evaluators

CONTACTS AND LOCATIONS:
Overall Officials: Georgi Petkov, Study Director — BTL Industries Ltd.